CLINICAL TRIAL: NCT00954954
Title: Outcomes After Standard and High-Flexion Posterior Stabilized Rotating-Platform Mobile-Bearing Total Knee Arthroplasty: A Prospective Randomized Comparative Study
Brief Title: Outcomes After Standard and High-Flexion Posterior Stabilized Rotating-Platform Mobile-Bearing Total Knee Arthroplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Myung Chul Lee / Professor, Seoul National University Hospital Department of Orthopaedic Surgery
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SNUHOSKNEE01-RPRPF
Record Dates: First submitted 2009-08-05; First posted 2009-08-07 (Estimated); Last update posted 2009-08-07 (Estimated); Status verified 2009-08

CONDITIONS: Osteoarthritis, Knee
Keywords: Arthroplasty; Replacement; Knee; Range of Motion
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard (Active Comparator): Knees that will be implanted with standard posterior stabilized RP-MB knee prostheses
  Interventions: Device: Standard PS RP-MB (P.F.C Sigma Rotating Platform knee)
- High-flexion (Active Comparator): Knees that will be implanted with high-flexion posterior stabilized RP-MB knee prostheses
  Interventions: Device: High-flexion PS RP-MB (P.F.C Sigma Rotating Platform Flex)

INTERVENTIONS:
Device: Standard PS RP-MB (P.F.C Sigma Rotating Platform knee) — Comparison of different types of knee prosthesis
  Other Names: P.F.C Sigma Rotating Platform knee
  Arms: Standard
Device: High-flexion PS RP-MB (P.F.C Sigma Rotating Platform Flex) — Comparison of different types of knee prosthesis
  Other Names: P.F.C Sigma Rotating Platform Flex
  Arms: High-flexion

SUMMARY:
The aim of this prospective study is to compare the clinical and radiographic outcomes of standard and high-flexion posterior stabilized (PS) rotating-platform mobile-bearing (RP-MB) total knee arthroplasty. The investigators hypothesize that total knee arthroplasty performed with a high-flexion PS RP-MB design would improve range of motion, and that this would be reflected by a better clinical outcome and greater patient satisfaction.

DETAILED DESCRIPTION:
A high-flexion, PS RP-MB prosthesis was designed to improve range of motion after total knee arthroplasty without compromising the theoretical advantages of the standard PS RP-MB system. To date, no study has prospectively compared the clinical and radiographic results of standard and high-flexion PS RP-MB designs.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of primary osteoarthritis of knee
* A candidate for total knee replacement arthroplasty

Exclusion Criteria:

* A diagnosis other than primary osteoarthritis
* A history of previous open knee surgery

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2006-10; Primary Completion 2007-06 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Range of knee motion, knee scores, patients' abilities to perform deep knee flexion related activities, patient satisfaction and radiographic indices were measured. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Myung Chul Lee, MD, PhD, Study Chair — Seoul National University Hospital Department of Orthopaedic Surgery
Locations (1):
- Seoul National University Hospital Department of Orthopaedic Surgery, Seoul, 28, Yongeon-Dong, Jongno-Gu, South Korea